CLINICAL TRIAL: NCT00499798
Title: Temozolomide Induced Changes in Semen/Sperm Analysis in Men With Newly Diagnosed, Progressive or Recurrent Primary Malignant Brain Tumors
Brief Title: Changes in Semen or Sperm Caused by Temozolomide in Patients With Newly Diagnosed, Progressive, or Recurrent Primary Malignant Brain Tumors
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000553297; CCCWFU-97404; CCCWFU-BG04-308
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2013-07

CONDITIONS: Brain and Central Nervous System Tumors; Chemotherapeutic Agent Toxicity; Infertility
Keywords: infertility; chemotherapeutic agent toxicity; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult giant cell glioblastoma; adult gliosarcoma; adult pilocytic astrocytoma; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult ependymoblastoma; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic meningioma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult papillary meningioma; adult grade I meningioma; adult grade II meningioma; adult grade III meningioma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult pineoblastoma; adult pineocytoma; adult mixed glioma; recurrent adult brain tumor; adult subependymal giant cell astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Infertility; Astrocytoma; Glioblastoma; Gliosarcoma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Medulloblastoma; Ependymoma; Glioma, Subependymal; Meningioma; Oligodendroglioma; Pinealoma; Glioma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients on temozolimide for brain cancer

SUMMARY:
RATIONALE: Learning whether temozolomide changes semen or sperm in patients with brain tumors may help doctors learn about the long-term effects of treatment and plan the best treatment.

PURPOSE: This clinical trial is studying changes in semen or sperm caused by temozolomide in patients with newly diagnosed, progressive, or recurrent primary malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess if temozolomide induces any changes in standard semen or sperm analysis parameters (i.e., volume, viscosity, pH, forward progression, total count, total motile count, motility, presence of round cells, agglutination, and morphology) in patients with newly diagnosed, recurrent, or progressive primary malignant brain tumors.

OUTLINE: This is a pilot study.

During treatment with temozolomide, patients undergo semen or sperm sample collection at baseline, 3 months, and 6 months for semen analysis. Samples are analyzed for volume, viscosity, pH, forward progression, total count, total motile count, motility, presence of round cells, agglutination, and morphology.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary malignant brain tumor

  * Newly diagnosed, progressive, or recurrent disease
  * May have received prior radiotherapy with or without chemotherapy
  * Scheduled to begin single-agent temozolomide chemotherapy
* Must be able to ejaculate

  * Must abstain from ejaculating (e.g., not have sex or masturbate) for 2-7 days prior to study
* No known abnormal sperm motility and/or morphology

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients recieving temozolimide for malignant brain tumor
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2004-08; Primary Completion 2009-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
assess any changes in standard semen/sperm analysis parameters | 6 months
  assess if Temozolomide induces any changes in standard semen/sperm analysis parameters (volume, viscosity, pH, forward progression, total count, total motile count, motility, presence of round cells, agglutination, and morphology)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J. Lesser, MD, Study Chair — Wake Forest University Health Sciences; Robert T. Blackwood, PA-S, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States